CLINICAL TRIAL: NCT00498810
Title: COMplete Versus PArtial Open inCisional Hernia Repair (COMPAC-TRIAL)
Acronym: COMPAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: patients had to be converted to the other study arm
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Frederik Berrevoet, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/241
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: complete repair
Procedure: partial repair of the abdominal wall

SUMMARY:
To compare the complete repair of the abdominal wall at the level of the former incision with only a partial repair at the level of the hernia in patients with an incisional hernia after median laparotomy in a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or his/her legal representative
* Incisional hernia requiring elective surgical repair

Exclusion Criteria:

* No written informed consent
* Emergency surgery (incarcerated hernia)
* All incisional or parastomal hernias not originating at the midline
* All recurrent hernias
* All patients with mesh placed intra-abdominally during surgery have to be withdrawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
recurrence rate | 1 year

SECONDARY OUTCOMES:
Perioperative morbidity rate
Postoperative pain
Long term complication rate
Recurrence rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be